CLINICAL TRIAL: NCT00316082
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial to Evaluate the Efficacy and Safety of Saxagliptin as Monotherapy With Titration in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control With Diet and Exercise
Brief Title: Study of BMS-477118 as Monotherapy With Titration in Subjects With Type 2 Diabetes Who Are Not Controlled With Diet and Exercise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV181-038
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Results first posted 2009-09-25 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — saxagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Saxagliptin 2.5 mg QAM (A) (Experimental): PLUS open-label metformin (as needed as rescue medication)
  Interventions: Drug: Saxagliptin; Drug: metformin
- Saxagliptin 2.5 mg titrated to 5 mg QAM (B) (Experimental): PLUS open-label metformin (as needed as rescue medication)
  Interventions: Drug: Saxagliptin; Drug: metformin
- Saxagliptin 5 mg QAM (C) (Experimental): PLUS open-label metformin (as needed as rescue medication)
  Interventions: Drug: Saxagliptin; Drug: metformin
- Saxagliptin 5 mg QPM (D) (Experimental): PLUS open-label metformin (as needed as rescue medication)
  Interventions: Drug: Saxagliptin; Drug: metformin
- Placebo (E) (Placebo Comparator): PLUS open-label metformin (as needed as rescue medication)
  Interventions: Drug: Placebo; Drug: metformin

INTERVENTIONS:
Drug: Saxagliptin — Coated tablets, Oral, 2.5 mg, QAM, Daily (6 months ST, 12 months LT)
  Other Names: BMS-477118
  Arms: Saxagliptin 2.5 mg QAM (A)
Drug: Saxagliptin — Coated tablets, Oral, 2.5 mg titrated to 5mg, QAM, Daily (6 months ST, 12 months LT)
  Other Names: BMS-477118
  Arms: Saxagliptin 2.5 mg titrated to 5 mg QAM (B)
Drug: Saxagliptin — Coated tablets, Oral, 5mg, QAM, Daily, (6 months ST, 12 months LT)
  Other Names: BMS-477118
  Arms: Saxagliptin 5 mg QAM (C)
Drug: Saxagliptin — Coated tablets, Oral, 5mg QPM, Daily (6 months ST, 12 months LT)
  Other Names: BMS-477118
  Arms: Saxagliptin 5 mg QPM (D)
Drug: Placebo — Coated tablets, Oral, 0mg, Daily (6 months ST, 12 months LT)
  Arms: Placebo (E)
Drug: metformin — Tablets, Oral, 500-2000 mg, as needed (12 months LT)

SUMMARY:
The purpose of this trial is to understand if saxagliptin is more effective than placebo as a treatment for type 2 diabetic subjects who are not controlled with diet and exercise

DETAILED DESCRIPTION:
All subjects will participate in a lead-in period, and qualifying subjects will continue into a short-term randomized treatment period. Subjects who complete the short-term period will be eligible to enter the long term extension period. Also, subjects in the short-term period who have an elevated blood sugar that requires additional medication for blood sugar control will be eligible to enter the long-term treatment extension period where they will receive metformin (rescue medication) added onto their blinded study medication

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Inadequate blood sugar control

Exclusion Criteria:

* Previous treatment for diabetes
* Current treatment with other medications to lower blood sugar
* Major heart, liver or kidney problems
* Women who are pregnant or breastfeeding

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2006-06; Primary Completion 2007-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (70):
- United States (51):
  - Tomac, Inc., Columbiana, Alabama
  - Winston Technology, Inc., Haleyville, Alabama
  - Clinical Reseacrh Advantage/ Brown Family Medicine, Mesa, Arizona
  - Strategos Medical Group, Bakersfield, California
  - Providence Clinical Research, Burbank, California
  - Rx For Life, Inc, Cudahy, California
  - Medical Group Of Encino, Encino, California
  - Southland Clinical Research Center, Inc., Fountain Valley, California
  - Valley Research, Fresno, California
  - Diabetes Medical Center Of California, Northridge, California
  - In Private Prictice Clinic, Pico Rivera, California
  - San Jose Clinical Research, Inc., San Jose, California
  - Central Florida Clinical Trials, Inc., Altamonte Springs, Florida
  - Accelovance, Melbourne, Florida
  - University Family Healthcare, Pa, Sarasota, Florida
  - Premier Healthcare, St. Petersburg, Florida
  - Pinnacle Medical Research, Overland Park, Kansas
  - Kansas City University Of Medicine And Biosciences, Kansas City, Missouri
  - Primary Care Physicians, Pc, Wentzville, Missouri
  - Physicians Research Center, Toms River, New Jersey
  - Hudson Valley Clinical Research Center, Kingston, New York
  - Neem Research Group Of Charlotte, Charlotte, North Carolina
  - Diabetes Center- East Carolina University, Greenville, North Carolina
  - Crescent Medical Research, Salisbury, North Carolina
  - Community Health Care, Inc., Barberton, Ohio
  - Clinical Research Limited, Canton, Ohio
  - Wells Institute For Health Awareness, Kettering, Ohio
  - Clinical Research Source, Inc, Perrysburg, Ohio
  - Accelovance, Oklahoma City, Oklahoma
  - Integris Family Care South, Oklahoma City, Oklahoma
  - The Office Of Patricia Buchanan, Eugene, Oregon
  - Cumberland Valley Endocrinology Center, Llc, Carlisle, Pennsylvania
  - Fleetwood Clinical Research, Fleetwood, Pennsylvania
  - Banksville Medical, Pc, Pittsburgh, Pennsylvania
  - Biomedical Research Associates, Llc, Shippensburg, Pennsylvania
  - Middle Tyger Family Medicine, Duncan, South Carolina
  - Southeastern Research Assoc, Taylors, South Carolina
  - Versoza & Ungab Internal Medicine Associates, Bartlett, Tennessee
  - Collierville Medical Specialist, Collierville, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Med-South Research, Memphis, Tennessee
  - Southwind Medical Specialist, Memphis, Tennessee
  - Precision Family Medicine, Carrollton, Texas
  - Alpha Therapy Research Center, Corpus Christi, Texas
  - Village Family Practice, Houston, Texas
  - Texas Center For Drug Development, P.A., Houston, Texas
  - Abbott Clinical Research Group, Inc, San Antonio, Texas
  - Taylor/Wade Medical, Bountiful, Utah
  - Optimum Clinical Research, Salt Lake City, Utah
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Spokane Internal Medicine, Spokane, Washington
- India (7):
  - Local Institution, Manipal, Karnataka
  - Local Institution, Kochi, Kerala
  - Local Institution, Attavar, Mangalore
  - Local Institution, Sarita Vihar, New Delhi
  - Local Institution, Bangalore
  - Local Institution, Mumbai
  - Local Institution, Nagpur
- Russia (7):
  - Local Institution, Moscov
  - Local Institution, Moscow
  - Local Institution, Nizhny Novgorod
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Smolensk
  - Local Institution, Volgograd
- Taiwan (5):
  - Local Institution, Changhua
  - Local Institution, Kaohsiung County
  - Local Institution, Taichung
  - Local Institution, Taipei
  - Local Institution, Tao-Yuan County

REFERENCES:
- [Derived] Perl S, Cook W, Wei C, Iqbal N, Hirshberg B. Saxagliptin Efficacy and Safety in Patients With Type 2 Diabetes and Moderate Renal Impairment. Diabetes Ther. 2016 Sep;7(3):527-35. doi: 10.1007/s13300-016-0184-9. Epub 2016 Jul 11. PMID 27402391
- [Derived] Bonora E, Bryzinski B, Hirshberg B, Cook W. A post hoc analysis of saxagliptin efficacy and safety in patients with type 2 diabetes stratified by UKPDS 10-year cardiovascular risk score. Nutr Metab Cardiovasc Dis. 2016 May;26(5):374-9. doi: 10.1016/j.numecd.2015.11.004. Epub 2015 Dec 1. PMID 27033025
- [Derived] Frederich R, McNeill R, Berglind N, Fleming D, Chen R. The efficacy and safety of the dipeptidyl peptidase-4 inhibitor saxagliptin in treatment-naive patients with type 2 diabetes mellitus: a randomized controlled trial. Diabetol Metab Syndr. 2012 Jul 24;4(1):36. doi: 10.1186/1758-5996-4-36. PMID 22828124

RESULTS

PARTICIPANT FLOW:
Groups:
- Saxagliptin 2.5 mg Once in the Morning (QAM): The Saxagliptin 2.5 mg QAM group includes data from subjects randomized to receive administration of blinded Saxagliptin 2.5 mg oral tablets QAM daily.
- Saxagliptin 5 mg QAM: The Saxagliptin 5 mg QAM group includes data from subjects randomized to receive administration of blinded Saxagliptin 5 mg oral tablets QAM daily.
- Saxagliptin 2.5/5 mg QAM: The Saxagliptin 2.5/5 mg QAM group includes data from subjects randomized to receive administration of blinded Saxagliptin 2.5 mg oral tablets QAM daily, with possible titration to 5 mg oral tablets QAM.
- Saxagliptin 5 mg Once in the Evening (QPM): The Saxagliptin 5 mg QPM group includes data from subjects randomized to receive administration of blinded Saxagliptin 5 mg oral tablets QPM daily.
- Placebo: The Placebo group includes data from subjects randomized to receive administration of placebo oral tablets daily.
Period: Overall Study
Arm/Group | Saxagliptin 2.5 mg Once in the Morning (QAM) | Saxagliptin 5 mg QAM | Saxagliptin 2.5/5 mg QAM | Saxagliptin 5 mg Once in the Evening (QPM) | Placebo
Started | 74 | 74 | 71 | 72 | 74
Completed Study Without Being Rescued | 25 | 35 | 29 | 27 | 31
Completed | 41 | 52 | 44 | 46 | 48
Not Completed | 33 | 22 | 27 | 26 | 26
Not completed — Lack of Efficacy | 2 | 3 | 3 | 4 | 6
Not completed — Withdrawal of Consent by Subject | 10 | 8 | 2 | 9 | 5
Not completed — Lost to Follow-up | 7 | 6 | 7 | 8 | 6
Not completed — Poor/noncompliance | 6 | 1 | 4 | 1 | 4
Not completed — Adverse Event | 4 | 2 | 5 | 1 | 3
Not completed — Subject no longer meets study criteria | 3 | 1 | 2 | 2 | 1
Not completed — Physician Decision | 1 | 1 | 2 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 0 | 0
Not completed — Administrative reason by sponsor | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 2.5 mg Once in the Morning (QAM) | Saxagliptin 5 mg QAM | Saxagliptin 2.5/5 mg QAM | Saxagliptin 5 mg Once in the Evening (QPM) | Placebo | Total
Number analyzed (Participants) | 74 | 74 | 71 | 72 | 74 | 365
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.24 (10.44) | 54.66 (9.71) | 54.28 (10.93) | 55.11 (10.35) | 55.57 (10.32) | 54.98 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 36 | 34 | 39 | 39 | 197
  Male | 25 | 38 | 37 | 33 | 35 | 168

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1 (A1C) at Week 24
Description: Mean change from baseline in A1C at Week 24, adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis of change from baseline to Week 24 Last Observation Carried Forward (LOCF), participants must have had a baseline and at least 1 post-baseline measurement. If participant received rescue medication, measurement must have been taken before rescue.
Measure: Mean (Standard Error); unit: percent
Groups:
- Saxagliptin 2.5 mg QAM: The Saxagliptin 2.5 mg QAM group includes data from subjects randomized to receive administration of blinded Saxagliptin 2.5 mg oral tablets QAM daily.
Arm/Group | Saxagliptin 2.5 mg QAM | Saxagliptin 5 mg QAM | Saxagliptin 2.5/5 mg QAM | Placebo
Number analyzed (Participants) | 67 | 69 | 69 | 68
percent
  Baseline Mean | 8.04 (0.105) | 7.93 (0.106) | 8.02 (0.131) | 7.79 (0.112)
  Week 24 Mean | 7.30 (0.106) | 7.27 (0.129) | 7.37 (0.137) | 7.57 (0.141)
  Adjusted Mean Change from Baseline | -0.71 (0.103) | -0.66 (0.102) | -0.63 (0.102) | -0.26 (0.103)

2. Secondary Outcome: Change From Baseline in A1C at Week 24 - Saxagliptin 5 mg QPM
Description: Mean change from baseline in A1C at Week 24, adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis of change from baseline to Week 24 LOCF, participants must have had a baseline and at least 1 post-baseline measurement. If a participant received rescue medication, then that measurement must have been taken before rescue.
Measure: Mean (Standard Error); unit: percent
Groups:
- Saxagliptin 5 mg QPM: The Saxagliptin 5 mg QPM group includes data from subjects randomized to receive administration of blinded Saxagliptin 5 mg oral tablets QPM daily.
Arm/Group | Saxagliptin 5 mg QPM | Placebo
Number analyzed (Participants) | 70 | 68
percent
  Baseline Mean | 7.88 (0.111) | 7.79 (0.112)
  Week 24 Mean | 7.29 (0.124) | 7.57 (0.141)
  Adjusted Mean Change from Baseline | -0.61 (0.101) | -0.26 (0.103)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Mean change from baseline in FPG at Week 24, adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg Once in the Morning (QAM) | Saxagliptin 5 mg QAM | Saxagliptin 2.5/5 mg QAM | Saxagliptin 5 mg Once in the Evening (QPM) | Placebo
Number analyzed (Participants) | 70 | 71 | 71 | 71 | 71
mg/dL
  Baseline Mean | 156.6 (3.96) | 162.2 (4.24) | 170.6 (6.15) | 159.6 (5.32) | 158.6 (5.44)
  Week 24 Mean | 146.8 (3.79) | 151.3 (5.88) | 155.2 (5.88) | 152.4 (5.88) | 162.9 (6.28)
  Adjusted Mean Change from Baseline | -11.4 (4.50) | -10.7 (4.46) | -12.5 (4.48) | -7.9 (4.46) | 3.3 (4.46)

4. Secondary Outcome: Percentage of Participants Achieving A1C < 7% at Week 24
Description: Percentage of participants achieving A1C < 7%, the American Diabetes Association's defined goal for glycemia, at each dose of saxagliptin versus placebo at Week 24.
Time Frame: Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in the Week 24 LOCF analysis, participants must have had at least 1 post-baseline measurement. If a participant received rescue medication, then that measurement must have been taken before rescue.
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin 2.5 mg Once in the Morning (QAM) | Saxagliptin 5 mg QAM | Saxagliptin 2.5/5 mg QAM | Saxagliptin 5 mg Once in the Evening (QPM) | Placebo
Number analyzed (Participants) | 67 | 69 | 69 | 70 | 68
Percentage of participants | 35.8 | 44.9 | 43.5 | 38.6 | 35.3

5. Secondary Outcome: Changes From Baseline in Postprandial Glucose (PPG) Area Under the Curve (AUC) Response to an Oral Glucose Tolerance Test (OGTT) at Week 24
Description: Mean change from baseline for 0 to 180 minutes PPG AUC at Week 24, adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg*min/dL
Arm/Group | Saxagliptin 2.5 mg Once in the Morning (QAM) | Saxagliptin 5 mg QAM | Saxagliptin 2.5/5 mg QAM | Saxagliptin 5 mg Once in the Evening (QPM) | Placebo
Number analyzed (Participants) | 48 | 48 | 47 | 43 | 47
mg*min/dL
  Baseline Mean | 47432 (1496.6) | 50417 (1561.5) | 50032 (1684.7) | 47078 (1941.9) | 47640 (1759.7)
  Week 24 Mean | 39798 (1347.0) | 41562 (1489.3) | 41745 (1739.2) | 41530 (1962.7) | 44861 (1854.7)
  Adjusted Mean Change from Baseline | -8014 (1246.9) | -8218 (1249.1) | -7781 (1261.0) | -6048 (1318.2) | -3088 (1259.7)

ADVERSE EVENTS:
Arm/Group | Placebo | Saxagliptin 2.5/5 mg QAM | Saxagliptin 2.5 mg QAM | Saxagliptin 5 mg QAM | Saxagliptin 5 mg QPM
Serious Adverse Events (participants affected / at risk) | 5/74 | 7/71 | 7/74 | 8/74 | 4/72
Other Adverse Events (participants affected / at risk) | 22/74 | 30/71 | 32/74 | 33/74 | 29/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=74) | Saxagliptin 2.5/5 mg QAM (N=71) | Saxagliptin 2.5 mg QAM (N=74) | Saxagliptin 5 mg QAM (N=74) | Saxagliptin 5 mg QPM (N=72)
RETINAL DETACHMENT (Eye disorders) | 0 | 0 | 0 | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
ANGINA UNSTABLE (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
COR PULMONALE ACUTE (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
ARTERIAL DISORDER (Vascular disorders) | 0 | 0 | 0 | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
RECTAL POLYP (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
FOOD POISONING (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
INFECTED BITES (Infections and infestations) | 0 | 1 | 0 | 0 | 0
PNEUMOCOCCAL SEPSIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
INTERTRIGO (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 1
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
CHEST PAIN (General disorders) | 0 | 1 | 1 | 0 | 0
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
HEPATIC CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=74) | Saxagliptin 2.5/5 mg QAM (N=71) | Saxagliptin 2.5 mg QAM (N=74) | Saxagliptin 5 mg QAM (N=74) | Saxagliptin 5 mg QPM (N=72)
HYPERTENSION (Vascular disorders) | 1 | 4 | 3 | 3 | 0
HEADACHE (Nervous system disorders) | 3 | 2 | 4 | 5 | 2
NAUSEA (Gastrointestinal disorders) | 1 | 4 | 4 | 2 | 3
DIARRHOEA (Gastrointestinal disorders) | 1 | 1 | 7 | 4 | 4
DYSPEPSIA (Gastrointestinal disorders) | 0 | 4 | 3 | 2 | 0
RHINITIS (Infections and infestations) | 1 | 4 | 0 | 1 | 0
SINUSITIS (Infections and infestations) | 3 | 5 | 5 | 3 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 3 | 1 | 5 | 1
NASOPHARYNGITIS (Infections and infestations) | 3 | 3 | 3 | 4 | 5
URINARY TRACT INFECTION (Infections and infestations) | 2 | 3 | 4 | 3 | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 11 | 11 | 10 | 11
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 4 | 3 | 5 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 1 | 5
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2 | 3 | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3 | 4 | 2
ASTHENIA (General disorders) | 3 | 4 | 0 | 1 | 2
OEDEMA PERIPHERAL (General disorders) | 3 | 2 | 5 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.